CLINICAL TRIAL: NCT04422236
Title: A Post-market, Observational Registry With the easyEndoTM Universal Linear Cutting Stapler in Laparoscopic Bariatric Surgery
Acronym: STAP-Delta
Status: Active, not recruiting | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: DM-Delta-01
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Roux-en-Y Gastric Bypass; Gastrectomy; Mini Gastric Bypass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients eligible for laparoscopic bariatric surgery
  Interventions: Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical)

INTERVENTIONS:
Device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) — Investigational device: easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical). Device for creation of anastomoses during laparoscopic bariatric surgery, manufactured by Ezisurg Medical.

SUMMARY:
The purpose of this observational registry is to evaluate the safety and performance of the easyEndoTM Universal Linear Cutting Stapler and reloads from Ezisurg Medical when used to create anastomoses during laparoscopic bariatric surgery. The goal of the study will be achieved by assessing the device performance and by reporting of peri- and postoperative complications in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age at registry entry.
* Patient and investigator signed and dated the informed consent form prior to the index-procedure.
* Patient has a BMI ≥ 35 kg/m2, with one or more related co-morbidities.
* Patient has a BMI ≥ 40 kg/m2.
* Patient is eligible for laparoscopic bariatric surgery.

Exclusion Criteria:

* Patient is unable / unwilling to provide informed consent.
* Patient has a history of bariatric surgery.
* Patient is unable to comply with the registry protocol or proposed follow-up visits.
* Patient has a contra-indication for laparoscopic bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients eligible for laparoscopic bariatric surgery. This registry will collect data from 200 laparoscopic bariatric procedures in which anastomoses are created with the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | At index procedure
  Conversion rate, number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | At discharge, up to 1 week
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | Follow-up 1: 3 weeks after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | Follow-up 2: 8 weeks after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | Follow-up 3: 6 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | Follow-up 4: 12 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | Follow-up 5: 18 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.
To evaluate the safety of the easyEndoTM Universal Linear Cutting Stapler and reloads (Ezisurg Medical) in laparoscopic bariatric surgery. | Follow-up 6: 24 months after the procedure
  Number of re-interventions and number of participants with (serious) adverse events ≥ grade II Clavien-Dindo.

SECONDARY OUTCOMES:
Device performance | At index procedure
  Number of procedures with technical success defined as bariatric surgery as intended, without technical difficulties and without conversion to open laparotomy.
Device performance | At index procedure
  Assessment of device performance (e.g. sharpness of the blade, staple-line formation, etc.).
Clinical efficacy | Follow-up 1: 3 weeks after the procedure
  Weight loss
Clinical efficacy | Follow-up 2: 8 weeks after the procedure
  Weight loss
Clinical efficacy | Follow-up 3: 6 months after the procedure
  Weight loss
Clinical efficacy | Follow-up 4: 12 months after the procedure
  Weight loss
Clinical efficacy | Follow-up 5: 18 months after the procedure
  Weight loss
Clinical efficacy | Follow-up 6: 24 months after the procedure
  Weight loss
Clinical efficacy | Follow-up 4: 12 months after the procedure
  Comorbidity
Clinical efficacy | Follow-up 6: 24 months after the procedure
  Comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Bart Smet, Dr., Principal Investigator — AZ Delta vzw
Locations (1):
- AZ Delta vzw, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No